CLINICAL TRIAL: NCT03955107
Title: The Effect of Continuous Glucose Monitoring on Glycemic Control and Pregnancy Outcomes in Gestational Diabetes Mellitus：A Randomized Controlled Trial.
Brief Title: The Effect of Continuous Glucose Monitoring on Glycemic Control and Pregnancy Outcomes in Gestational Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yufan Wang, Director of endocrinology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTCCR-2018BP02
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Gestational Diabetes; Continuous Glucose Monitoring
Keywords: gestational diabetes; continuous glucose monitoring; glycemic Control
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: This is a open-label, randomized controlled trial. The investigators plan to recruit 154 women with gestational diabetes at 24-28 weeks gestation. 77 subjects (Group 1) will be selected to undergo CGM every 4 weeks and another 77 subjects will be recruited to undergo usual antenatal care ,and last month undergo CGMS (Group 2).
  The primary outcomes will be time in range of glycaemic control in the third trimester. The investigators also plan to assess changes to management made by the endocrinologist based on the additional information on glycemic control obtained from professional CGM use. The investigators also plan to compare hypoglycaemia and hyperglycaemia detection rates using the CGMS and fingerstick methods of glucose evaluation. Written and informed consent will be obtained in accordance with the principles of the Helsinki Declaration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous Glucose Monitoring System (Other)
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Patients in the intervention group will receive Continuous Glucose Monitoring(CGMS) every 4 weeks since diagnosed with GDM，and the control grouponly once receive CGMS during the last month and have management adjusted based on the CGMS readings Other Name: iPro, Medtronic

SUMMARY:
The purpose of this study is to determine if Continuous glucose monitoring improves glycemic control and pregnancy outcomes of Gestational Diabetes Mellitus

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as any degree of glucose intolerance that is first identified during pregnancy, excluding diabetic patients diagnosed before pregnancy. The purpose of this study is to determine if Continuous glucose monitoring improves glycemic control and pregnancy outcomes of Gestational Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* women with gestational diabetes
* 18-45 years old
* 24-28 weeks gestation of pregnancy
* singleton pregnancy
* BMI≥18kg/m2

Exclusion Criteria:

* pregestational type 1 or 2 diabetes mellitus
* aged <18 or >45 years
* BMI<18kg/m2
* multiple pregnancy
* Cushing's syndrome/ using exogenous steroids
* chronic infection ( HIV, Hepatitis B/C, Tuberculosis)
* any active chronic systemic disease ( except essential hypertension)
* Severe liver and kidney dysfunction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
time in range at Week 8 after enrollment | at Week 8 after enrollment
  time in range of CGMS at Week 8 after enrollment

SECONDARY OUTCOMES:
the level of HbA1c before delivery | 37 weeks of gestation
  the level of HbA1c before delivery in two groups
the incidence of hypoglycemic events | 14 weeks
  the incidence of hypoglycemic events (blood glucose <3.3mmol/L, with or without hypoglycemic symptoms) during the follow-up period of patients in the two groups
adverse pregnancy outcomes | 3 month
  adverse pregnancy outcomes (preterm, macrosomia, greater than gestational age, less than gestational age, compound end point (birth injury, neonatal hypoglycemia, hyperbilirubinemia, apgar score < 7 within 5 minutes of birth, neonatal phototherapy, neonatal respiratory distress syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai Jiao Tong University 100 Haining Road,Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No